CLINICAL TRIAL: NCT07103148
Title: A Parallel Group, Phase III Randomized, Modified Double-blind, Active Controlled Study to Investigate the Immunogenicity and Safety of vYF Compared to Licensed YF Vaccines in Pediatric Population Aged 9 Months to 5 Years of Age
Brief Title: A Phase III Control Study of the Safety and Immunogenicity of vYF in Pediatric Population
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VYF04; VYF04 (Other: Sanofi Identifier); U1111-1300-4387 (Other: WHO ICTRP)
Record Dates: First submitted 2025-07-07; First posted 2025-08-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Yellow Fever Immunization
Keywords: Yellow fever
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Sponsor, Investigators, Study staff who conduct the safety assessment and the participant' parent(s) / LAR(s) will not know which study intervention is administered.
  * Only the study staff who prepare and administer the study interventions and are not involved with the safety evaluation will know which study intervention is administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1 (9-24 months) (Experimental): Primary vaccination phase: 1 injection of vYF vaccine at Day 1 Booster phase: 1 injection of vYF vaccine at Year 3 (in a subset)
  Interventions: Biological: Yellow fever vaccine (live)
- Group 2 (9-24 months) (Active Comparator): Primary vaccination phase: 1 injection of Stamaril vaccine at Day 1 Booster phase: 1 injection of Stamaril vaccine at Year 3 (in a subset)
  Interventions: Biological: Yellow fever vaccine (live)
- Group 3 (9-24 months) (Active Comparator): Primary vaccination phase: 1 injection of YF-VAX vaccine at Day 1 Booster phase: 1 injection of YF-VAX vaccine at Year 3 (in a subset)
  Interventions: Biological: Yellow fever vaccine (live)
- Group 4 (2-5 years) (Experimental): Primary vaccination phase: 1 injection of vYF vaccine at Day 1
  Interventions: Biological: Yellow fever vaccine (live)
- Group 5 (2-5 years) (Active Comparator): Primary vaccination phase: 1 injection of Stamaril vaccine at Day 1
  Interventions: Biological: Yellow fever vaccine (live)
- Group 6 (2-5 years) (Active Comparator): Primary vaccination phase: 1 injection of YF-VAX vaccine at Day 1
  Interventions: Biological: Yellow fever vaccine (live)
- Group 7 (approximately 11-15 months) (Experimental): Primary vaccination phase: 1 injection of MMR vaccine at Day 1 in a cohort of 11 to 15 months of age vaccinated with vYF
  Interventions: Biological: Yellow fever vaccine (live); Biological: Measles, combinations with mumps and rubella, live attenuated

INTERVENTIONS:
Biological: Yellow fever vaccine (live) — Powder and diluent for suspension for injection Subcutaneous
  Other Names: vYF vaccine
  Arms: Group 1 (9-24 months); Group 4 (2-5 years); Group 7 (approximately 11-15 months)
Biological: Yellow fever vaccine (live) — Powder and diluent for suspension for injection Subcutaneous
  Other Names: Stamaril vaccine
  Arms: Group 2 (9-24 months); Group 5 (2-5 years)
Biological: Yellow fever vaccine (live) — Powder and diluent for suspension for injection Subcutaneous
  Other Names: YF-VAX vaccine
  Arms: Group 3 (9-24 months); Group 6 (2-5 years)
Biological: Measles, combinations with mumps and rubella, live attenuated — Powder, lyophilized, for suspension for reconstitution Subcutaneous or intermuscular
  Other Names: MMR II vaccine
  Arms: Group 7 (approximately 11-15 months)

SUMMARY:
The purpose of this study is to determine whether vYF (investigational vaccine) is safe and can help the body to develop antibodies (immunogenicity) compared with Stamaril vaccine and YF-VAX vaccine (both licensed vaccines) and when they are co-administered with Measles Mumps Rubella (MMR) vaccines in infants aged 11-15 months.

Number of Participants:

A total of 2440 participants is planned to be enrolled in VYF04 study.

Study Arms and Duration:

Eligible participants will be randomized in 2 independent groups (9-24 months, 2-5 years) to receive 1 dose of either vYF or Stamaril or YF-VAX in a 2:1:1 ratio within each age group. An additional group with participants of 11-15 months of age will also receive at the same vaccination visit vYF and a single dose of MMR vaccine.

For the 2nd step (YF booster vaccine administration in a subset), at the Year (Y) 3 visit, a subset of 120 participants of the 9-24 months of age group who did receive a YF vaccine on Day(D) 01 will be invited to join a booster dose assessment (booster dose administered after the Y3 visit blood sample has been taken). Participants aged 11 to 15 months at the time of the concomitant administration of vYF and MMR will not be eligible for receiving a booster dose.

The duration of each participation will be approximately 3 years for all participants (including participants co-administered on D01 with vYF and MMR), and 6 more months post-booster dose administration for the participants enrolled in the booster subset.

DETAILED DESCRIPTION:
The duration of each participant's participation will be up to approximately 3 years (not including booster phase in a subset)

The Phase III VYF04 is the first study to be carried out with the investigational vYF in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 months to 5 years on the day of inclusion*

  * "9 months to 5 years" means from the day of the 9th month after birth to the day before the 6th year birthday
* Aged 11 to 15 months* on the day of inclusion for participants enrolled in the MMR co-administration group

  * "11 to 15 months" means from the day of the 11th month after birth to the day before the 16th month birthday
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* For infants*, born after a gestation period of 27 through 36 weeks and medically stable as assessed by the investigator, based on the following definition: "Medically stable" refers to the condition of premature infants who do not require significant medical support or ongoing management for debilitating disease and who have demonstrated a clinical course of sustained recovery by the time they receive the first dose of study intervention

  * Infants aged 9 months to 11 months up to the day before the 12th month birthday
* Participant and parent/LAR are able to attend all scheduled visits and to comply with all study procedures
* ICF has been signed and dated by the parent(s) or other LAR (and by an independent witness if required by local regulations)

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy irradiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known history of FV infection
* Known systemic hypersensitivity to any of the study intervention components, eggs or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Chronic illness* that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion , including malignancy, such as leukemia, or lymphoma

  *Chronic illness may include, but is not limited to, cardiac disorders, renal disorders, auto-immune disorders, diabetes, psychiatric disorders or chronic infection
* History of central nervous system disorder or disease, including seizures and febrile seizures
* Receipt of any vaccine in the 4 weeks preceding the study intervention administration or planned receipt of any vaccine in the 4 weeks following the study intervention administration. Vaccine to be administered as part of the National Immunization Schedule will be postponed after the D29 visit
* Previous vaccination against a FV disease at any time including YF with an investigational or marketed vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 6 months
* Administration of any anti-viral within 2 months preceding the study intervention administration and up to the 6 weeks following the study intervention administration
* For participants enrolled in the MMR co-administration group: previous vaccination against measles, measles/mumps/rubella
* For participants enrolled in the MMR co-administration group: history of measles, mumps, rubella confirmed either clinically, serologically, or microbiologically
* Known history or laboratory evidence of HIV infection
* Known history of hepatitis B or hepatitis C seropositivity
* Personal or family history of thymic pathology (thymoma, thymectomy, or myasthenia)
* Participation at the time of study enrollment (or in the 4 weeks preceding the study intervention administration) or planned participation during the first year of the 3-year follow-up in another clinical study investigating a vaccine, drug, medical device, or medical procedure. Enrollment in another study after the first 6 months of follow-up is permitted, assuming it does not exclude participation in this study.
* In an emergency setting, or hospitalized involuntary
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study

Ages: 9 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2440 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2030-03-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with seroconversion to YF virus after 1 dose of vYF compared to seroconversion after 1 dose of the Stamaril in YF-naive participants (9-24 months) | At Day 29, 28 days post-vaccination (on Day 01) with vYF or Stamaril
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in NAb titers as compared to the pre-vaccination value
Percentage of participants with seroconversion to YF virus after 1 dose of vYF compared to seroconversion after 1 dose of the YF-VAX in YF-naive participants (9-24 months) | At Day 29, 28 days post-vaccination (on Day 01) with vYF or YF-VAX
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in NAb titers as compared to the pre-vaccination value
Percentage of participants with seroconversion to YF virus after 1 dose of vYF compared to seroconversion after 1 dose of the Stamaril in YF-naive participants (2-5 years) | At Day 29, 28 days post-vaccination (on Day 01) with vYF or Stamaril
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in NAb titers as compared to the pre-vaccination value
Percentage of participants with seroconversion to YF virus after 1 dose of vYF compared to seroconversion after 1 dose of the YF-VAX in YF-naive participants (2-5 years) | At Day 29, 28 days post-vaccination (on Day 01) with vYF or YF-VAX
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in NAb titers as compared to the pre-vaccination value

SECONDARY OUTCOMES:
Percentage of participants, by age group, with seroconversion to YF virus in all investigational vaccine groups before (Day 01) and after investigational vaccine administration at various timepoints | At Day 01 and at Day 11 (in a subset), Day 15 (in a subset), Day 29, Month 6, and yearly from Year 1 to Year 3
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in NAb titers as compared to the pre-vaccination value
Percentage of participants, by age group, with seroprotection to YF virus in all investigational vaccine groups before (Day 01) and after investigational vaccine administration at various timepoints | At Day 01 and at Day 11 (in a subset), Day 15 (in a subset), Day 29, Month 6, and yearly from Year 1 to Year 3
  Seroprotection is defined as NAb titers ≥ 10 (1/dil) at the corresponding timepoint
Geometric Mean Titers (GMTs) of neutralizing antibodies against YF virus in all investigational vaccine groups, by age group, before (Day 01) and after investigational vaccine administration at various timepoints | At Day 01 and at Day 11 (in a subset), Day 15 (in a subset), Day 29, Month 6, and yearly from Year 1 to Year 3
  Antibody titers are expressed as geometric mean titers
Geometric Mean Titers Ratio (GMTRs) of neutralizing antibodies against YF virus in all investigational vaccine groups, by age group, before (Day 01) and after investigational vaccine administration at various timepoints | GMTRs Day 11/Day 01 (subset only), Day 15/ D01 (subset only), Day 29/Day 01, Month 6/Day 01, Year 1/Month 6, Year 2/Year 1, Year 3/Year 2
  At Day 01 and at Day 11 (in a subset), Day 15 (in a subset), Day 29, Month 6, and yearly from Year 1 to Year 3
Percentage of participants with seroconversion to YF virus in all investigational vaccine groups 28 days after the co-administration of vYF with measlescontaining vaccine in the MMR group and at successive timepoints | 28 days after the coadministration of MMR with vYF At Month 6 and yearly from Year 1 to Year 3
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in NAb titers as compared to the prevaccination value
Percentage of participants with seroprotection to YF virus in all investigational vaccine groups 28 days after the co-administration of vYF with measlescontaining vaccine in the MMR group and at successive timepoints | 28 days after the coadministration of MMR with vYF At Month 6 and yearly from Year 1 to Year 3
  Seroprotection is defined as NAb titers ≥ 10 (1/dil) at the corresponding timepoint
GMTs of neutralizing antibodies against YF virus in all investigational vaccine groups 28 days after the co-administration of vYF with measlescontaining vaccine in the MMR group and at successive timepoints | 28 days after the coadministration of MMR with vYF At Month 6 and yearly from Year 1 to Year 3
  Antibody titers are expressed as geometric mean titers
GMTRs of neutralizing antibodies against YF virus in all investigational vaccine groups 28 days after the co-administration of vYF with measlescontaining vaccine in the MMR group and at successive timepoints | 28 days after the coadministration of MMR with vYF At Month 6 and yearly from Year 1 to Year 3
  GMTRs Day 29/Day 01, Month 6/Day 01, Year 1/Month 6, Year 2/Year 1, Year 3/Year 2
Percentage of participants, by age group, with seroconversion to YF virus in all investigational vaccine groups before (Day 01) and after investigational vaccine administration at various timepoints | Before and 28 days after the coadministration of MMR with vYF
  Seroconversion is defined for measles, mumps and rubella respectively in participants seronegative at baseline as an antibody titer reaching the following thresholds for seropositivity:
  * Anti-measles antibody concentrations ≥ 255 mIU/mL
  * Anti-mumps antibody concentrations ≥ 10 (AbU)/mL
  * Anti-rubella antibody concentrations ≥ 10 IU/mL
Percentage of participants with seroprotection to MMR before and 28 days after the coadministration of MMR with vYF in the MMR group | Before and 28 days after the coadministration of MMR with vYF
GMTs of neutralizing antibodies against MMR virus before and 28 days after the coadministration of MMR with vYF in the MMR group | Before and 28 days after the coadministration of MMR with vYF
  Antibody titers are expressed as geometric mean titers
GMTRs of neutralizing antibodies against MMR virus before and 28 days after the coadministration of MMR with vYF in the MMR group | Before and 28 days after the coadministration of MMR with vYF
  GMTRs Day 29/Day 01
Percentage of participants with seroconversion to YF virus before the booster dose administration at Y3, then 10 days and 28 days after a vYF booster dose in the booster subset | At Day 11 and Day 29 after booster dose
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in NAb titers as compared to the prevaccination value
Percentage of participants with seroprotection to YF virus before the booster dose administration at Y3, then 10 days and 28 days after a vYF booster dose in the booster subset | At Day 11 and Day 29 after booster dose
  Seroprotection is defined as NAb titers ≥ 10 (1/dil) at the corresponding timepoint
GMTs of neutralizing antibodies against YF virus before the booster dose administration at Y3, then 10 days and 28 days after a vYF booster dose in the booster subset | At Day 11 and Day 29 after booster dose
  Antibody titers are expressed as geometric mean titers
GMTRs of neutralizing antibodies against YF virus before the booster dose administration at Y3, then 10 days and 28 days after a vYF booster dose in the booster subset | At Day 11 and Day 29 after booster dose
  GMTRs Day 11/D01 and Day 29/Day 01
Percentage of participants with seroconversion to YF up to Day 29 will be described depending on the FV status at baseline (YF, Dengue, Zika) by age group | Up to Day 29
  YF and Zika NAbs will be measured using a qualified MN assay Quantitation of human IgG antibodies against dengue virus (DENV) nonstructural protein 1 (NS1) in human sera will be determined using a qualified ELISA assay. Seroconversion is defined as a 4-fold increase in NAb titers as compared to the prevaccination value
Percentage of participants with seroprotection to YF up to Day 29 will be described depending on the FV status at baseline (YF, Dengue, Zika) by age group | Up to Day 29
  Seroprotection is defined as NAb titers ≥ 10 (1/dil) at the corresponding timepoint
GMTs of neutralizing antibodies against YF up to Day 29 will be described depending on the FV status at baseline (YF, Dengue, Zika) by age group | Up to Day 29
  Antibody titers are expressed as geometric mean titers
GMTRs of neutralizing antibodies against YF up to Day 29 will be described depending on the FV status at baseline (YF, Dengue, Zika) by age group | Up to Day 29
  GMTRs Day 29/Day 01
Number of participants with immediate adverse events | Within 30 minutes after each vaccination
  Immediate adverse events are any unsolicited systemic adverse events reported in the 30 minutes after vaccination
Number of participants with solicited injection site reactions | Within 7 days after each vaccination
  Solicited injection site reactions:
  * for participants < 24 months include: injection site tenderness, injection site erythema, injection site swelling
  * for participants aged ≥ 2 years and < 5 years include: injection site pain, injection site erythema and injection site swelling
Number of participants with solicited systemic reactions | Within 14 days after each vaccination
  Solicited systemic reactions:
  * for participants < 24 months include: fever, vomiting, crying abnormal, drowsiness, appetite lost, irritability
  * for participants aged ≥ 2 years and < 5 years include: fever, headache, fatigue and myalgia
Number of participants with unsolicited adverse events (AEs) | Within 28 days after each vaccination
  Unsolicited (spontaneously reported) AEs, not fulfilling criteria for solicited adverse reactions
Number of participants with medically attended adverse events (MAAEs) | From Day 01 to Day 29
  MAAEs will be collected as part of the unsolicited AEs
Number of participants with serious adverse events (SAEs) and adverse events of special interest (AESIs) | From Day 01 to Month 6 and from Year 3 to Year 3 + 6 Months for the booster subset
  SAEs and AESIs
Hematology in a subset of participants 9-24 months of age and in a subset of participants aged 2-5 years | At Day 01 and at Day 05
  Blood samples will be taken for the determination of hematology
Biochemistry in a subset of participants 9-24 months of age and in a subset of participants aged 2-5 years | At Day 01 and at Day 05
  Blood samples will be taken for the determination of biochemistry
YF vaccinal viremia in each vaccine groups (vYF, Stamaril and YF-VAX) in a subset of participants 9-24 months of age | At Day 01 and at Day 05
  YF vaccinal viremia will be measured by YF-specific quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay

CONTACTS AND LOCATIONS:
Locations (8):
- Honduras (3):
  - Investigational Site Number : 3400001, San Pedro Sula
  - Investigational Site Number : 3400002, Tegucigalpa
  - Investigational Site Number : 3400003, Tegucigalpa
- Mexico (5):
  - Investigational Site Number : 4840007, Torreón, Coahuila
  - Investigational Site Number : 4840013, Cuernavaca, Morelos
  - Investigational Site Number : 4840015, Tizimín, Yucatán
  - Investigational Site Number : 4840009, Chihuahua City
  - Investigational Site Number : 4840005, Ecatepec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VYF04 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26787&tenant=MT_SNY_9011